CLINICAL TRIAL: NCT04882527
Title: Modulating Prospective Memory in Older Adults With Noninvasive Brain Stimulation
Brief Title: Modulating Prospective Memory in Older Adults With Non-invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-01599
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- anodal stimulation of the rIFL (Experimental): Anodal stimulation over the right inferior frontal lobe
  Interventions: Device: Non-invasive brain stimulation
- cathodal stimulation of the rIFL (Experimental): Cathodal stimulation over the right inferior frontal lobe
  Interventions: Device: Non-invasive brain stimulation
- anodal stimulation of the lIFL (Experimental): Anodal stimulation over the left inferior frontal lobe
  Interventions: Device: Non-invasive brain stimulation
- cathodal stimulation of the lIFL (Experimental): Cathodal stimulation over the left inferior frontal lobe
  Interventions: Device: Non-invasive brain stimulation
- anodal stimulation of the rSPL (Experimental): Anodal stimulation over the right superior parietal lobe
  Interventions: Device: Non-invasive brain stimulation
- cathodal stimulation of the rSPL (Experimental): Cathodal stimulation over the right superior parietal lobe
  Interventions: Device: Non-invasive brain stimulation
- sham stimulation (Sham Comparator): Sham stimulation over either of the three real stimulation areas
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Non-invasive brain stimulation — Stimulation will be applied once per subject with one mA for 20 minutes over either the left inferior frontal lobe, the right inferior frontal lobe or the right superior parietal lobe.
  Other Names: high-definition transcranial direct current stimulation; HD-tDCS; Soterix medical
  Arms: anodal stimulation of the lIFL; anodal stimulation of the rIFL; anodal stimulation of the rSPL; cathodal stimulation of the lIFL; cathodal stimulation of the rIFL; cathodal stimulation of the rSPL
Device: Sham stimulation — The electrode positions and the attachment procedures correspond to those of real tDCS but the electrical current will only be ramped up to 1 mA and switched off completely after 30 s of stimulation.
  Arms: sham stimulation

SUMMARY:
Prospective memory is the ability to remember to carry out intentions with a certain delay (e.g. remember to buy stamps when passing a postal office). Prospective memory tasks require a large degree of self-initiated retrieval and in the absence of a prompt to recall, people must 'remember to remember' by their own volition. Thus, prospective memory is a challenge - especially in old age with increasing health-related prospective memory demands.

Previous studies reported links between neural activity in specific brain regions and prospective memory performance. Yet, the mere occurrence of a change in brain activity in concomitance with performance of a behavioral task is not sufficient to confirm a causal relationship between the two phenomena. Therefore, this study aims to apply non-invasive brain stimulation to facilitate or inhibit activity in different brain regions presumed to be functionally associated with prospective memory. Additional to the prospective memory tasks, the investigators will implement control tasks (i.e., attention) to assess whether stimulation will specifically enhance prospective memory performance or whether other cognitive functions will be modulated additionally.

It is hypothesized that stimulation will lead to changes in prospective memory functioning. Further, the investigators expect that facilitation of attentional processes might be linked to prospective memory improvements.

DETAILED DESCRIPTION:
This study aims to modulate neural activity in the left and right inferior frontal lobe as well as in the right superior parietal lobe via high-definition transcranial direct current stimulation (HD-tDCS) in older adults. There is evidence from functional magnetic resonance imaging (fMRI) studies that these areas are involved in prospective memory performance in younger and older adults but a causal relation between activity in these areas and responses in prospective memory tasks has not been established so far.

A double blind, sham-controlled, parallel group design will be applied. Healthy older adults (n=105) will participate in two separate sessions: During the first baseline session, no stimulation is applied. For the second session, participants will then be randomly assigned to one of seven experimental groups (cathodal vs. anodal right inferior frontal lobe (rIFL); cathodal vs. anodal left inferior frontal lobe (lIFL); cathodal vs. anodal right superior parietal lobe (rSPL); or sham). Real stimulation will be applied during 20 minutes with one Milliamp (mA). In case of sham stimulation (i.e., control intervention), the electrode positions and the attachment procedures correspond to those of real tDCS but the electrical current will only be ramped up to one mA and switched off completely after 30 s of stimulation.

The primary objective of this study is the modulation of prospective memory performance in a computer-based task via tDCS. Further, this study aims to clarify the role of attentional control for prospective memory performance, as both processes seem to recruit similar neural structures. Additionally, naturalistic and self-rated prospective memory performance will be assessed.

It is hypothesized that stimulation of the right inferior frontal lobe will lead to changes in prospective memory performance and attentional processes. Whether cathodal or anodal stimulation will enhance performance is not clear yet, since previous fMRI studies were inconsistent about activity changes in older adults. Further, the investigators expect that anodal stimulation of the left inferior frontal cortex may lead to faster responses to prospective memory stimuli, whereas cathodal stimulation of the same area may lead to prolonged reaction times. It is hypothesized that attentional control will not be affected by stimulation of the left inferior frontal lobe. Finally, the investigators expect that anodal stimulation of the right superior parietal cortex will lead to better prospective memory and attentional control performance, whereas cathodal stimulation will have detrimental effects on both functions.

ELIGIBILITY:
Inclusion Criteria:

* No cognitive impairments
* Fluent in German
* Right-handed
* Normal or corrected-to-normal vision
* Non-smokers
* Written informed consent

Exclusion Criteria:

* Current/lifetime severe psychiatric or neurological disorder
* Metal implants in the head area
* Psychotropic medication
* Dermatosis
* Current/lifetime alcohol abuse
* Magnetisable implants

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female participants will be equally distributed between groups.
Enrollment: 106 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Prospective memory performance | During both sessions (for stimulation session: during intervention), fixed to 14 minutes
  Assessed with a computer task. Number of correct answers given to prospective memory stimuli.
  Change from baseline to intervention session, difference between intervention groups.
Prospective memory reaction time | During both sessions (for stimulation session: during intervention), fixed to 14 minutes
  Assessed with a computer task. Reaction times of answers given to prospective memory stimuli.
  Change from baseline to intervention session, difference between intervention groups.
Executive controlling functioning | During both sessions (for stimulation session: during intervention), task fixed to 6 minutes
  Assessed with a computer task (ANT - Attentional Network Task). Interference between answers given to congruent and incongruent stimuli.
  Change from baseline to intervention session, difference between intervention groups.
Flexibility performance | During both sessions (for stimulation session: directly after intervention), 3 minutes
  Assessed with a computer task (TAP- Test of Attentional Performance). Number of correct answers.
  Change from baseline to intervention session, difference between intervention groups.
Inhibition errors | During both sessions (for stimulation session: directly after intervention), 2 minutes
  Assessed with a computer task (Test of Attentional Performance). Sum of incorrect responses to no-go stimuli.
  Change from baseline to intervention session, difference between intervention groups.
Divided attention misses | During both sessions (for stimulation session: directly after intervention), 3 minutes 30 seconds
  Assessed with a computer task (TAP - Test of Attentional Performance). Sum of missed target stimuli.
  Change from baseline to intervention session, difference between intervention groups.
Flexibility reaction-time | During both sessions (for stimulation session: directly after intervention), 3 minutes
  Assessed with a computer task (TAP - Test of Attentional Performance). Mean/ median of reactions times of correct responses.
  Change from baseline to intervention session, difference between intervention groups.
Inhibition reaction time | During both sessions (for stimulation session: directly after intervention), 2 minutes
  Assessed with a go/no-go computer task (TAP -Test of Attentional Performance). Mean/ median of reactions times to correct responses.
  Change from baseline to intervention session, difference between intervention groups.
Divided attention reaction time | During both sessions (for stimulation session: directly after stimulation), 3 minutes 30 seconds
  Assessed with a computer-based task (Test of Attentional Performance). Median reaction time of correct answers.
  Change from baseline to intervention session, difference between intervention groups.

SECONDARY OUTCOMES:
Alerting network functioning | During both sessions (for stimulation session: during intervention), task fixed to 6 minutes
  Assessed with a computer task (ANT - Attentional Network Task). Contrasting reaction times of answers given to stimuli with alerting cues to those without alerting cues.
  Change from baseline to intervention session, difference between intervention groups.
Orienting network functioning | During both sessions (for stimulation session: during intervention), task fixed to 6 minutes
  Assessed with a computer task (ANT - Attentional Network Task). Contrasting reaction times of answers given to stimuli with reliable spatial cues to those without spatial cues.
  Change from baseline to intervention session, difference between intervention groups.
Ongoing-task performance | During both sessions (for stimulation session: during intervention), fixed to 14 minutes
  Assessed with a computer task. Number of correctly answered ongoing task stimuli in the course of the prospective memory task.
  Change from baseline to intervention session, difference between intervention groups.
Ongoing-task reaction time | During both sessions (for stimulation session: during intervention), fixed to 14 minutes
  Assessed with a computer task. Mean/median response time of correct ongoing task answers in the course of the prospective memory task.
  Change from baseline to intervention session, difference between intervention groups.
Ongoing-task intra-individual coefficient of variation | During both sessions (for stimulation session: during intervention), fixed to 14 minutes
  Assessed with a computer task. Variability of response times (i.e., within-person fluctuation in response latency) to ongoing task stimuli in the course of the prospective memory task.
  Change from baseline to intervention session, difference between intervention groups.

OTHER OUTCOMES:
Self-rated prospective memory | Only at baseline session, after computer-based tasks, 10 minutes
  Assessed with a questionnaire (PRMQ - Prospective Retrospective Memory Questionnaire).
  Comparison to performance in other tasks.
Self-rated metacognitive prospective memory | Only at stimulation session, after intervention, 10 minutes
  Assessed with a questionnaire (MPMI - Metacognitive Prospective Memory Inventory).
  Comparison to performance in other tasks.
Stimulation Side-Effects | Only at stimulation session, after intervention, 3 minutes
  Self-rating about adverse side effects during and after stimulation are assessed with a questionnaire.
Naturalistic prospective memory | 5 minutes per session; retrieval within five days after each session
  Assessed with a behavioral task. Number of correctly retrieved naturalistic prospective memory intentions.
  Change from baseline to intervention session, difference between intervention groups.
Inhibition intra-individual coefficient of variation | During both sessions (for stimulation session: directly after intervention), 2 minutes
  Assessed with a go/no-go computer task (TAP -Test of Attentional Performance). Variability of response times (i.e., within-person fluctuation in response latency) to go-stimuli.
  Change from baseline to intervention session, difference between intervention groups.
Flexibility intra-individual coefficient of variation | During both sessions (for stimulation session: directly after intervention), 3 minutes
  Assessed with flexibility computer task (TAP -Test of Attentional Performance). Variability of response times (i.e., within-person fluctuation in response latency).
  Change from baseline to intervention session, difference between intervention groups.
Divided attention intra-individual coefficient of variation | During both sessions (for stimulation session: directly after stimulation), 3 minutes 30 seconds
  Assessed with a computer-based task (Test of Attentional Performance). Variability of response times (i.e., within-person fluctuation in response latency).
  Change from baseline to intervention session, difference between intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Klöppel, Prof. Dr., Principal Investigator — University of Bern; Jessica Peter, PD Dr., Study Chair — University of Bern; Matthias Kliegel, Prof. Dr., Study Chair — University of Geneva; Nadine Schmidt, MSc., Study Chair — University of Bern
Locations (1):
- Universitätsklinik für Alterspsychiatrie und Psychotherapie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt N, Menendez-Granda M, Munger R, Reber TP, Bayen UJ, Gumusdagli FE, Hering A, Joly-Burra E, Kliegel M, Peter J. Modulating prospective memory and attentional control with high-definition transcranial current stimulation: Study protocol of a randomized, double-blind, and sham-controlled trial in healthy older adults. PLoS One. 2023 Aug 7;18(8):e0289532. doi: 10.1371/journal.pone.0289532. eCollection 2023. PMID 37549139